CLINICAL TRIAL: NCT02847130
Title: Use of Evidence-Based Supportive Care Clinical Practice Guidelines in Pediatric Oncology
Brief Title: Identifying, Understanding, and Overcoming Barriers to the Use of Clinical Practice Guidelines in Pediatric Oncology
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCL15N1CD; NCI-2016-00980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL15N1CD (Other: Children's Oncology Group); COG-ACCL15N1CD (Other: DCP); ACCL15N1CD (Other: CTEP); UG1CA189955 (NIH)
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-04

CONDITIONS: Acute Lymphoblastic Leukemia; B-Cell Non-Hodgkin Lymphoma; Childhood Acute Myeloid Leukemia; Childhood Burkitt Lymphoma; Childhood Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Recurrent Childhood Acute Lymphoblastic Leukemia
Keywords: Clinical practice guidelines; supportive care; pediatrics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell; Burkitt Lymphoma; Neoplasms; Hematologic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (chart review, focus group, interviews): AIM 1 (CHART REVIEW): Patients are separated for each CPG evaluated (fever and neutropenia [FN], chemotherapy induced nausea and vomiting [CINV], fertility preservation [FP]) and are randomly selected for medical chart review. Patients with eligible episodes of FN, CINV or FP within the health records are selected and have the data from their records abstracted and reviewed by COG for adherence to COG endorsed CPGs.
  AIM 2 (FOCUS GROUPS): Health care providers who provide direct care to pediatric oncology patients are identified and separated to participate in three types of focus groups: physician-only, non-physician, and mixed.
  AIM 3 (INTERVIEWS): Health care providers undergo one-on-one interviews consisting of think aloud technique (TAL) of cognitive interviewing.
  Interventions: Other: Informational Intervention; Other: Interview; Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Informational Intervention — Participate in focus group
Other: Interview — Undergo one-on-one interviews
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the use of clinical practice guidelines by pediatric oncology healthcare providers in order to identify, understand, and overcome barriers to them. The treatments for childhood cancers are intense and result in a high rate of symptoms which require support by healthcare providers. By reviewing patients' medical chart records, meeting in focus groups and in one-on-one interviews, healthcare providers may improve how clinical practice guidelines are used to support children undergoing cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the rate of adherence to selected Children's Oncology Group (COG)-endorsed supportive care clinical practice guidelines (CPG) recommendations at National Cancer Institute (NCI) Community Oncology Research Program (NCORP) sites. (Aim 1) II. To describe the possible influence of NCORP site size and the number of patients enrolled in COG studies per site on the delivery of CPG-consistent care. (Aim 1a) III. To describe the clinical outcome of episodes during which patients receive CPG-consistent or CPG-inconsistent care. (Aim 1b) IV. To describe facilitators of and barriers to the use of CPGs elicited via focus group interviews with a diverse set of potential users (physician, nurse, nurse practitioner and pharmacists) who provide pediatric cancer care at NCORP sites. (Aim 2) V. To improve how well CPG recommendations are understood by health care providers by refining the CPG recommendation format based on an iterative process of cognitive interviewing and formatting revisions. (Aim 3)

OUTLINE:

AIM 1 (CHART REVIEW): Patients are separated for each CPG evaluated (fever and neutropenia [FN], chemotherapy induced nausea and vomiting [CINV], fertility preservation [FP]) and are randomly selected for medical chart review. Patients with eligible episodes of FN, CINV or FP within the health records are selected and have the data from their records abstracted and reviewed by COG for adherence to COG endorsed CPGs.

AIM 2 (FOCUS GROUPS): Health care providers who provide direct care to pediatric oncology patients are identified and separated to participate in three types of focus groups: physician-only, non-physician, and mixed.

AIM 3 (INTERVIEWS): Health care providers undergo one-on-one interviews consisting of think aloud technique (TAL) of cognitive interviewing.

ELIGIBILITY:
Inclusion Criteria:

* Site willingness to participate in all 3 aims
* AIM 1 - ELIGIBILITY CRITERIA FOR INCLUSION IN RETROSPECTIVE CENTRALIZED CHART REVIEW
* Received care as an inpatient or outpatient at a participating COG NCORP site during the time period between January 1, 2014 and December 31, 2015
* Ever enrolled on any COG trial (episode does not have to occur while on trial and the COG trial may be therapeutic or non-therapeutic)
* Has at least one episode eligible for FN, CINV or FP review
* CPG-Specific Eligibility
* FN

  * Has any of the following diagnoses:

    * Newly diagnosed acute lymphoblastic leukemia
    * Relapsed acute lymphoblastic leukemia
    * Any acute myeloid leukemia
    * Burkitt's or mature B cell non-Hodgkin's lymphoma
    * Any myeloablative autologous or allogeneic hematopoietic stem cell transplantation
    * Developed FN at least once
* CINV

  * Diagnosis of cancer
  * Received moderately emetogenic chemotherapy as an inpatient
  * < 12 years of age at the start of a CINV episode and received highly emetogenic chemotherapy as an in-patient
* FP

  * Newly diagnosed cancer
  * >= 15 years of age at cancer diagnosis
* Note: a single patient may contribute data for multiple episodes
* AIM 2 AND AIM 3 INCLUSION CRITERIA
* Healthcare professional currently employed at a participating COG NCORP institution

  * Eligible healthcare providers include but are not limited to: physicians, nurses, nurse practitioners, pharmacists, social workers, dieticians, psychologists, and physical therapists/physiotherapists
* Provides direct care for children with cancer as part of current position at NCORP site

Exclusion Criteria:

* AIM 2 AND AIM 3 EXCLUSION CRITERIA
* Trainees are excluded
* Previous participation in this study either for Aim 2 or Aim 3
* Each health care provider can only be involved in one event (focus group or interview)

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients < 21 years old at cancer diagnosis who received care as an inpatient or outpatient at a participating COG NCORP site between January 1, 2014 and December 31, 2015
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The proportion of clinical practice guidelines (CPG)-consistent care of fever and neutropenia (FN) episodes | Care delivered from January 1, 2014 through December 31, 2015 will be evaluated
  FN will be identified by chart review. Outcome variable will be the binary endpoint of CPG-consistent versus (vs.) CPG inconsistent care for each FN episode.
The proportion of CPG-consistent care of chemotherapy induced nausea and vomiting (CINV) episodes | Care delivered from January 1, 2014 through December 31, 2015 will be evaluated
  CINV will be identified by chart review. Outcome variable will be the binary endpoint of CPG-consistent vs. CPG inconsistent care for each CINV episode (separately for high and moderate emetogenicity risk chemotherapy).
The proportion of CPG-consistent care of fertility preservation (FP) episodes | Care delivered from January 1, 2014 through December 31, 2015 will be evaluated
  FP will be identified by chart review. Outcome variable will be the binary endpoint of CPG-consistent vs. CPG inconsistent care for each FP episode.
Possible influence of National Cancer Institute Community Oncology Research Program site size (Aim 1a) | Care delivered from January 1, 2014 through December 31, 2015 will be evaluated
  Will be estimated and examined as fixed effect covariates in these generalized linear mixed effect models described above.
Key coding categories (Aim 2) | Data collected from March 28, 2017 through October 15, 2018 will be evaluated
  Will be identified by the Framework for Clinical Practice Guideline Implementability. Operational definitions of each category will be determined. The implementation barriers and facilitators identified by focus group members will be coded using these categories independently by two investigators. New categories and sub-categories will be used to code concepts that do not fall within the pre-determined categories. Themes of commonality will be sought especially within the newly developed categories that fall outside the framework adapted from Gagliardi et al. Facilitators of and barriers to CPG implementation will be described.
CPG format which is well understood by pediatric oncology healthcare providers (Aim 3) | Data collected from a minimum of 25 interviews starting from February 1, 2019 to the timepoint where a format that is well understood by participants is developed will be evaluated
  The issues identified via the interviews, changes made to the formatting, and rationale for the changes will be documented between each round in a tracking matrix. The proportion of interviewees who select the correct course of action when presented with four possible courses of action will be described for each iteration of the CPG format including the final version. Understanding is defined as the correct interpretation of the course of action recommended or suggested by a CPG.

CONTACTS AND LOCATIONS:
Overall Officials: L. Lee Dupuis, Principal Investigator — Children's Oncology Group
Locations (33):
- United States (31):
  - Kaiser Permanente-Oakland, Oakland, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Blank Children's Hospital, Des Moines, Iowa
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Sugalski AJ, Lo T, Beauchemin M, Grimes AC, Robinson PD, Walsh AM, Santesso N, Dang H, Fisher BT, Wrightson AR, Yu LC, Sung L, Dupuis LL. Facilitators and barriers to clinical practice guideline-consistent supportive care at pediatric oncology institutions: a Children's Oncology Group study. Implement Sci Commun. 2021 Sep 16;2(1):106. doi: 10.1186/s43058-021-00200-2. PMID 34530933